CLINICAL TRIAL: NCT05533723
Title: Comparison Between Endoscopic Epidural Neuroplasty and Percutaneous Epidural Neuroplasty With a Steering Catheter in Low Back and Radicular Pain
Brief Title: Comparison Between Endoscopic Epidural Neuroplasty and Percutaneous Epidural Neuroplasty in Low Back and Radicular Pain
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Bum Choi, professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-MDB-20-53
Record Dates: First submitted 2022-08-23; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain; Radiculopathy
MeSH Terms: conditions — Low Back Pain; Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Percutaneous epidural neuroplasty (PEN) group: Patients over 20 years of age with radiating pain in the lower back and legs who received PEN in patients who did not respond to medication and epidural nerve block treatment.
  Interventions: Procedure: Percutaneous epidural neuroplasty (PEN)
- Endoscopic epidural neuroplasty (EEN) group: Patients over 20 years of age with radiating pain in the lower back and legs who received EEN in patients who did not respond to medication and epidural nerve block treatment.
  Interventions: Procedure: Endoscopic epidural neuroplasty

INTERVENTIONS:
Procedure: Endoscopic epidural neuroplasty — EEN catheter, iDolphine S2 (Meta Biomed Co., Ltd, Osong, Korea) was placed in the epidural space through sacral hiatus. EEN was done on the target segments.
  During EEN, normal saline was infused into epidural space under epiduroscopic vision. Dexamethasone (5 mg), 0.3% mepivacaine 10 mL, and hyaluronidase (3000 IU) were injected through catheter at the target segments. Holmium-Yag laser was used to cut epidural fibrous bands and for coagulation of epidural bleeding.
  Other Names: Percutaneous epidural neuroplasty (PEN)
  Groups: Endoscopic epidural neuroplasty (EEN) group
Procedure: Percutaneous epidural neuroplasty (PEN) — PEN catheter, EDEN-CC (JMT, Yangju, Korea) was placed in the epidural space and neural foramen . PEN was done on the target segments. Dexamethasone (5 mg), 0.3% mepivacaine 10 ml, and hyaluronidase (3000 IU) were injected through the PEN catheter.
  Groups: Percutaneous epidural neuroplasty (PEN) group

SUMMARY:
PEN(percutaneous epidural neuroplasty) can be performed percutaneously, may be manipulated to mechanically break up adhesions by catheter, while various agents, such as anesthetics, corticosteroids, hyaluronidase, and hypertonic saline are injected. In endoscopic epidural neuroplasty (EEN), a flexible catheter is inserted into the sacral hiatus to precisely place the injection in the epidural space and onto the nerve root. Both EEN and PEN can eliminate the deleterious effects of scar formation, which can physically prevent the direct application of drugs to the nerves, and may provide pain relief in patients who have not responded to epidural blocks, physical therapy, or medication. In this study, visual analog scale (VAS) and Oswestry disability index (ODI) of patients with low back and radicular pain were compared in patients who had received EEN or PEN at 1 day, 1 month, and 6 months after EEN or PEN.

DETAILED DESCRIPTION:
Low back pain and lumbar radicular pain commonly occur in degenerative spondy-losis. Low back and radicular pain have many underlying causes, one of which is scar-ring in the epidural space, which can cause pain for many reasons. The nerves may be trapped by scars, while the congestive veins in the epidural space can become enlarged and exert pressure upon the nerves.

Percutaneous epidural neuroplasty (PEN) with a wire type catheter, first reported by Dr. Racz, has been widely practiced since 1989, and reduces pain by epidural adhesiolysis, epidural fibrosis and inflammation near the neural tissue.

The PEN procedure is used to dissolve some scar tissue around the entrapped nerves in the epidural space of the spine. PEN can be performed percutaneously, using a Racz catheter. The catheter may be manipulated to mechanically break up adhesions, while various agents, such as anesthetics, corticosteroids, hyaluronidase, and hypertonic saline are injected. In endoscopic epidural neuroplasty (EEN), a flexible catheter is inserted into the sacral hiatus to precisely place the injection in the epidural space and onto the nerve root. Both EEN and PEN can eliminate the deleterious effects of scar formation, which can physically prevent the direct application of drugs to the nerves, and may pro-vide pain relief in patients who have not responded to epidural blocks, physical therapy, or medication.

In this study, visual analog scale (VAS) and Oswestry disability index (ODI) of pa-tients with low back and radicular pain were compared in patients who had received EEN or PEN at 1 day, 1 month, and 6 months after EEN or PEN.

ELIGIBILITY:
Inclusion Criteria:

1. age over 20 years
2. low back or radicular pain in the low extremities
3. persistent low back or radicular pain

Exclusion Criteria:

1. systemic infection
2. skin infection at the injection site
3. uncontrolled diabetes mellitus
4. coagulation abnormalities
5. history of allergic reactions to local anesthetics or contrast agents

Age Groups: Child, Adult, Older Adult
Study Population: Patients who visited Ajou University Hospital pain clinic with back and radiating pain from 2016 to 2020
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 6 months after EEN or PEN
  11 points pain scale score from 0 to 10
Oswestry disability index | 6 months after EEN or PEN
  disability index from 0 to 100%

SECONDARY OUTCOMES:
weight | before EEN or PEN
  kg
height | before EEN or PEN
  m

CONTACTS AND LOCATIONS:
Overall Officials: Jong Bum Choi, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyunggi, South Korea

IPD SHARING:
Plan to Share IPD: No